CLINICAL TRIAL: NCT06782763
Title: A Randomized Controlled Study on the Efficacy and Safety of Task-activated rTMS in Improving Cognitive Function in Patients With Bipolar Disorder
Brief Title: Efficacy and Safety of Task-activated rTMS in Improving Cognitive Function in Patients With Bipolar Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIT20240151C
Record Dates: First submitted 2025-01-01; First posted 2025-01-20 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-12

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- rTMS active group and active cognitive training (Experimental): Receive 10 Hz, 20 minutes of active rTMS stimulation; 20 minutes of cognitive training at the same time
  Interventions: Device: Repetitive transcranial magnetic stimulation device
- rTMS active group and sham cognitive training (Sham Comparator): 10 Hz, 20 minutes of active rTMS stimulation; 20 minutes of perform simple judgment training at the same time
  Interventions: Device: Repetitive transcranial magnetic stimulation device
- rTMS sham group and active cognitive training (Sham Comparator): 10 Hz, 20 minutes of low-intensity rTMS stimulation; 20 minutes of cognitive training at the same time
  Interventions: Device: Repetitive transcranial magnetic stimulation device
- rTMS sham group and sham cognitive training (Sham Comparator): 10 Hz, 20 minutes of low-intensity rTMS stimulation; perform simple judgment training for 20 minutes at the same time
  Interventions: Device: Repetitive transcranial magnetic stimulation device

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation device — Activating neurons: rTMS can activate or inhibit neuronal activity in certain brain areas, changing the activity pattern of neural networks. Neuroplasticity: By changing the strength and connection mode of synapses, it promotes the plasticity of the nervous system, which helps treat neuropsychiatric diseases. Regulating neurotransmitters: rTMS can regulate the release of neurotransmitters, affect nerve conduction, and thus improve disease symptoms.
  Other Names: Cognitive training

SUMMARY:
1. To clarify the efficacy and safety of task-based repetitive transcranial magnetic stimulation (rTMS) on cognitive function in patients with stable bipolar disorder.
2. To analyze the therapeutic mechanism of transcranial magnetic stimulation based on magnetic resonance imaging and explore the abnormal regulation mechanism of cognitive neural circuits.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 14 to 45 years, right-handed;
2. Meet the diagnostic criteria for bipolar disorder in the stable remission period of the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5);
3. Stable medication treatment;
4. Clinical remission for more than three months, Young Mania Rating Scale (YMRS) ≤ 6 points Hamilton Depression Rating Scale 17 (HDRS 17) score ≤ 7 points;
5. Cognitive impairment on the Cognitive Deficit Questionnaire (PDQ) ≥ 17 points;
6. Fully understand the transcranial magnetic stimulation treatment, be willing to actively cooperate with the treatment, and sign the informed consent.

Exclusion Criteria:

1. Those with a history of severe physical illness or diseases that may affect the central nervous system (such as tumors, syphilis, etc.);
2. Those with neurological diseases or risk of epileptic seizures, such as previous craniocerebral diseases, head trauma, alcoholism, abnormal EEG, MRI evidence of abnormal brain structure, or a family history of epilepsy;
3. Those with contraindications to MRI scanning or transcranial magnetic stimulation treatment, such as those with metal or electronic devices in the body (metal foreign bodies in the brain, cochlear implants, pacemakers and stents);
4. Those at high risk of suicide, or those who have already committed suicide or serious self-harm and need emergency intervention;
5. Those who are pregnant, breastfeeding, or planning to become pregnant during the trial;
6. Those with color blindness or hearing impairment;
7. Those with a history of substance or alcohol abuse;
8. Other situations that the researcher determines are not suitable as research subjects.

Ages: 14 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 82 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
PDQ-21 | 0-5 days
  The Perceived Deficits Questionnaire-21 (PDQ-21) is a widely used self-report scale designed to assess cognitive dysfunction in individuals with various medical and psychiatric conditions. It is particularly valuable in conditions where cognitive impairment, such as problems with memory, attention, and executive functioning, significantly impacts daily life.Total scores range from 0 to 84, with higher scores indicating greater perceived cognitive impairment.

SECONDARY OUTCOMES:
brain imaging (MRI) | 0-5 days
  Functional and structural changes in brain imaging (MRI)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China